CLINICAL TRIAL: NCT06221020
Title: To Assess the Impact of the Enhanced Recovery After Surgery (ERAS) Consensus on the Effectiveness and Prognosis of Patients With Endoscopic Pituitary Tumor Surgery
Brief Title: To Assess the Impact of theERAS Consensus on Patients With Endoscopic Pituitary Tumor Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202300876B0A3
Record Dates: First submitted 2023-12-04; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Enhanced Recovery After Surgery; Pituitary Tumor; Postoperative Complications
Keywords: Enhanced Recovery After Surgery; Pituitary tumor; Anesthesia Safety; Postoperative Complications
MeSH Terms: conditions — Pituitary Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — pituitary tumor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ERAS: In the experimental group (Patients with ERAS), participants will undergo an assessment of the Enhanced Recovery After Surgery (ERAS) consensus items.
  The experimental group will complete all the items on the ERAS forms as far as possible. All groups will undergo our routine preoperative evaluation for pituitary tumor surgery, such as cardiopulmonary function, hormone testing, vision and visual field examination, etc. The care during hospitalization and surgery will be the same as previously for patients with pituitary tumors, and the post-discharge outpatient follow-up will also be the same as for patients who have undergone pituitary tumor surgery.
  Interventions: Diagnostic Test: Malnutrition Universal Screening Tool; Device: TIB Olfactory Test Device; Diagnostic Test: Apfel Score for Postoperative nausea and vomiting; Diagnostic Test: The American Society of Anesthesiologists (ASA) Physical Status Classification; Behavioral: Short Form-36; Behavioral: World Health Organization Quality of Life questionnaire (WHOQOL-BREF); Behavioral: BDI-II(Beck Depression Inventory-II); Behavioral: ERAS Patient Satisfaction Questionnaire(ERAS-PSQ); Behavioral: Quality of Recovery-40(QoR-40)
- Patients with Regular: In the control group (Patients with Regular), participants will only complete the routine items as before.
  All groups will undergo our routine preoperative evaluation for pituitary tumor surgery, such as cardiopulmonary function, hormone testing, vision and visual field examination, etc. The care during hospitalization and surgery will be the same as previously for patients with pituitary tumors, and the post-discharge outpatient follow-up will also be the same as for patients who have undergone pituitary tumor surgery.
  Interventions: Diagnostic Test: Malnutrition Universal Screening Tool; Device: TIB Olfactory Test Device; Diagnostic Test: Apfel Score for Postoperative nausea and vomiting; Diagnostic Test: The American Society of Anesthesiologists (ASA) Physical Status Classification; Behavioral: Short Form-36; Behavioral: World Health Organization Quality of Life questionnaire (WHOQOL-BREF); Behavioral: BDI-II(Beck Depression Inventory-II); Behavioral: ERAS Patient Satisfaction Questionnaire(ERAS-PSQ); Behavioral: Quality of Recovery-40(QoR-40)

INTERVENTIONS:
Diagnostic Test: Malnutrition Universal Screening Tool — The Malnutrition Universal Screening Tool (MUST) is a commonly used tool for assessing the nutritional status of adult patients. It is designed to identify early whether a patient is at risk of malnutrition or is already malnourished, enabling timely intervention and treatment. MUST includes three main assessment criteria:
  Body Mass Index (BMI):
  Degree of Weight Loss: This assesses the patient's weight change over the past three months, with grading based on the extent of weight loss.
  Effect of Illness on Dietary Intake: This evaluates the impact of illness on the patient's dietary intake, with grading based on the reduction in dietary intake.
  By combining the grades from these three assessment indicators, a final MUST score is obtained to determine the patient's nutritional status and level of risk. Based on the MUST score, patients can be categorized as low risk, medium risk, or high risk for malnutrition.
Device: TIB Olfactory Test Device — Olfactory testing is conducted on patients undergoing pituitary tumor surgery via nasal endoscopy using the TIB Olfactory Test Device (TIBSIT). This testing aims to compare olfactory (sense of smell) outcomes before and after the surgery. The olfactory tests are performed preoperatively and then again at the 3-month postoperative mark to assess any changes or impacts on the sense of smell due to the surgery.
Diagnostic Test: Apfel Score for Postoperative nausea and vomiting — Nausea and Vomiting Risk Scale: Apfel Score
  Risk Factors: Female; Smoking habit; History of postoperative nausea and vomiting or motion sickness; Use of opioid painkillers post-surgery (Each risk factor scores 1 point; minimum score is 0; maximum score is 4)
  Score Probability of Postoperative Nausea and Vomiting
  0 - 10%
  1. - 21%
  2. - 39%
  3. - 61%
  4. - 79%
Diagnostic Test: The American Society of Anesthesiologists (ASA) Physical Status Classification — ASA I: A normal, healthy patient with no systemic disease. ASA II: A patient with mild systemic disease. ASA III: A patient with severe systemic disease that limits activity but is not incapacitating.
  ASA IV: A patient with severe systemic disease that is a constant threat to life.
  ASA V: A moribund patient not expected to survive without the operation. This project involves collecting data from adult patients aged 20 to 75 years old who are classified as ASA I to III grade.
Behavioral: Short Form-36 — The Short Form-36 (SF-36) is a widely used health assessment tool, extensively applied in both research and clinical practice. It is a concise yet comprehensive questionnaire designed to evaluate individuals' health status and quality of life. The SF-36 covers eight different dimensions of health, including physical functioning, bodily pain, general health, vitality, social functioning, emotional health, mental health, and health change. Each dimension is assessed through a series of questions that address aspects such as an individual's capabilities in daily life, symptoms, and emotional states. The SF-36 allows healthcare professionals and researchers to gain insights into a person's health and quality of life across these varied aspects. Additionally, SF-36 has undergone extensive testing and validation, proving to have good reliability and validity.
Behavioral: World Health Organization Quality of Life questionnaire (WHOQOL-BREF) — The World Health Organization Quality of Life questionnaire (WHOQOL-BREF) is a health-related quality of life assessment tool developed by the World Health Organization (WHO). It is designed to evaluate an individual's satisfaction with their life and overall health status. The WHOQOL-BREF is a condensed version of the original WHOQOL-100 questionnaire, intended to reduce the time required to complete it and enhance its applicability.
Behavioral: BDI-II(Beck Depression Inventory-II) — The BDI-II consists of 21 questions that assess the degree of depression by asking respondents about various depressive symptoms they have experienced. These symptoms include sadness, insomnia or oversleeping, changes in appetite, self-blame, self-disdain, loss of interest in daily activities, and more. Each question has four possible response options, allowing respondents to choose the answer that best fits their feelings.
  Scoring on the BDI-II ranges from 0 to 63, with higher scores indicating more severe depression. Based on the scores, the severity of a respondent's depression can be classified into different levels, ranging from mild to severe. The purpose of using this scale is to help healthcare professionals assess a patient's depressive symptoms, monitor changes in condition, and evaluate the effectiveness of treatments.
Behavioral: ERAS Patient Satisfaction Questionnaire(ERAS-PSQ) — The ERAS Patient Satisfaction Questionnaire (ERAS-PSQ) is a satisfaction survey specifically designed for patients who have undergone treatment following the Enhanced Recovery After Surgery (ERAS) protocols. This questionnaire aims to evaluate the patients' satisfaction and experience with the ERAS approach. Typically, it includes questions about various aspects of their treatment and care, such as pain management, the recovery process, the quality of nursing care, and communication with the medical team. The ERAS-PSQ is an important tool for assessing how well the ERAS protocols are received by patients and for identifying areas for improvement in patient care within the ERAS framework.
Behavioral: Quality of Recovery-40(QoR-40) — The Quality of Recovery-40 (QoR-40) is a widely used questionnaire designed to assess the quality of recovery after surgery. It comprises 40 questions that cover both physical and psychological aspects of a patient's recovery, such as pain, nausea, anxiety, dietary habits, and social functioning. The QoR-40 provides a comprehensive view of a patient's postoperative recovery, encompassing a range of factors crucial to understanding the effectiveness of surgical procedures and the overall patient experience during the recovery phase. This tool is instrumental in evaluating and improving post-surgical care and patient outcomes.

SUMMARY:
The goal of this observational study is to evaluate the effectiveness and impact of Enhanced Recovery After Surgery (ERAS) on patients with pituitary gland tumors.

DETAILED DESCRIPTION:
The goal of this observational study is to evaluate the effectiveness and impact of Enhanced Recovery After Surgery (ERAS) on patients with pituitary gland tumors. This study is particularly significant as ERAS has been a prominent focus in international medical treatment, emphasizing improved patient recovery and safety. The main questions it aims to answer are:

How does ERAS affect the effectiveness and prognosis of patients with pituitary gland tumors? Which specific inspection and evaluation items within the ERAS protocol genuinely assist patients? Participants in this study will undergo various ERAS protocols, including pre-operative to post-operative rehabilitation measures, pain management, surgical techniques, and early resumption of eating and activities. This comprehensive approach is designed to reduce complications, shorten hospital stays, and speed up patient recovery.

Additionally, this study will conduct a thorough statistical analysis to determine which aspects of the ERAS protocol are most beneficial. By comparing the outcomes of patients undergoing the ERAS protocol with those who do not, researchers aim to understand better the balance between ERAS and the Choosing Wisely initiative, which advocates for reducing unnecessary medical interventions.

This research is crucial in advancing medical knowledge and practice, particularly in managing pituitary gland tumors, and contributes to the broader goals of enhancing medical quality and patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pituitary tumors
* To sign a written informed consent form

Exclusion Criteria:

* Diagnosed with other malignant tumors
* Severe infections, such as osteomyelitis, acute inflammation at the affected site, or open wounds at the treatment area
* Pregnant women
* Coagulation disorders or those taking anticoagulant medication
* Other central nervous system disorders, alcohol addiction, other addictive drugs, or mental illness that may affect clinical assessment
* Deemed unsuitable for surgical treatment or unable to comply with clinical evaluation upon assessment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pituitary tumors, primarily benign growths, develop in the pituitary gland situated in the sellar region. This gland plays a pivotal role in regulating vital body functions including growth, metabolism, and various hormonal functions. As these tumors enlarge, they may press on adjacent areas and impair the gland's functions, leading to symptoms like headaches, vision issues, and hormonal imbalances.
  The principal treatment for pituitary tumors is surgery, aiming to excise the tumor from the brain's base. This procedure alleviates pressure on the pituitary gland and nearby structures, aiming to reinstate the gland's normal functionality.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Surgical complications | three months after operation
  any complications associated with this operation
Postoperative pain assessment | During the hospitalization period, up to 24 weeks
  describe postoperative Visual analogue scale (VAS) for pain assessment; the minimum value is 0 (no pain) and maximum value is 10 (most pain)
Postoperative vomiting assessment | During the postoperative period, up to 7 days
  describe postoperative vomiting status; 0=no; 1=mild, 2=moderate, 3=severe
Postoperative nausea assessment | During the postoperative period, up to 7 days
  describe postoperative nausea status; 0=no; 1=mild, 2=moderate, 3=severe
Reoperation during hospitalization | During the hospitalization period, the time from the first surgery to the reoperation is related to this surgical procedure, assessment up to 12 weeks.
  Reoperation during hospitalization related to this surgery.
Length of hospital stay | The duration from the day of admission to the day of discharge, which is associated with this surgical procedure, assessment up to 12 weeks.
  days of hospitalization related to this surgery.
Readmission within 30 days | within 30 days related to this surgery.
  Readmission within 30 days related to this surgery.

SECONDARY OUTCOMES:
Psychological stress- BDI-II | through study completion, an average of 1 year
  using Beck Depression Inventory-II, assessment of Psychological stress before and after surgery
Psychological stress- QoR-40 | through study completion, an average of 1 year
  using Quality of Recovery-40, assessment of Psychological stress before and after surgery
Quality of life: Short Form-36 | through study completion, an average of 1 year
  assessment of Quality of life before and after surgery
Quality of life: WHOQOL-BREF | through study completion, an average of 1 year
  assessment of Quality of life before and after surgery
ERAS Patient Satisfaction Questionnaire | through study completion, an average of 1 year
  assessment of Patient Satisfaction for this study

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chen Wang, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan